CLINICAL TRIAL: NCT06704906
Title: Assess Clinical and Radiographic Outcomes of VIPER PRIME/Expedium Spine System and Fibergraft BG Putty
Brief Title: Adult Patient Outcomes After Spine Surgery With Fibergraft BG Putty/Viper Prime
Status: Recruiting | Type: Observational
Sponsor: Nitin Agarwal (Other)
Collaborators: DePuy Synthes (Industry)
Responsible Party: Sponsor-Investigator, Nitin Agarwal, Associate Professor, Neurosurgery, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: STUDY24040006
Record Dates: First submitted 2024-10-28; First posted 2024-11-26 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Spondylolisthesis, Lumbar Region; Spinal Trauma With Neurological Deficit; Degeneration of Lumbar Intervertebral Disc
MeSH Terms: conditions — Spondylolisthesis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Use of Viper Prime/Expedium system with Fibergraft BG Putty — Patients who require spine surgery under standard of care and meet the inclusion and exclusion criteria identified, will be recruited from clinic. Consent for participation in study will be signed at the same time as consent for surgery. All PROMs and scans will be done as standard of care and data will be obtained through chart review for this study.

SUMMARY:
The Viper Prime/Expedium spine systems are intended to provide immobilization and stabilization of spinal segments in skeletally mature patients as an adjunct to fusion in the treatment of acute and chronic instabilities or deformities of the thoracolumbar and sacral spine. The Fibergraft Bioactive Glass (BG) is engineered to mimic the body's natural bone healing process. While previous studies have compared the use of Viper prime/Expedium spine system in minimally invasive and open surgeries, these studies did not specifically study the clinical and radiographic outcomes of patients who have received these implants in addition to Fibergraft. We aim to recruit patients with degenerative disc disease, spondylolisthesis, trauma, and/or pseudarthrosis who require spine surgery under standard of care and use these implants. We will then follow these patients for a duration of two years to report their clinical and radiographic outcomes to determine fusion, complication rate, and revision surgeries if any.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Have a radiograph-based diagnosis of degenerative disc disease, spondylolisthesis, spinal trauma (i.e., fracture or dislocation), spinal stenosis, or deformity (i.e., scoliosis, kyphosis, and/or lordosis), spinal tumor, or pseudoarthrosis/failed fusion.
3. Pathology of the thoracolumbar or sacral spine.
4. Patients requiring fusion of 1-3 levels
5. Patients receiving the surgery/devices as standard of care prescribed by the treating physician.

Exclusion Criteria:

1. Patients < 18 years
2. Patients with a cervical spine pathology
3. Patients with spinal tumors
4. Patients with bone density (DEXA) scores < 2.0 will be excluded.
5. Current smokers and patients who quit smoking within 6 weeks prior to presentation will be excluded.
6. Patients with a BMI > 40kg/m2
7. Patients requiring fusion for more than 3 levels will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with spinal conditions mentioned in inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Fusion | 2 years (At baseline, postoperatively at 6 weeks, 3 months, 6 months, 12 months, and 24 months)
  We will assess fusion with regular x-rays and CT scans at 1 and 2-year postoperatively.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | 2 years (At baseline, postoperatively at 6 weeks, 3 months, 6 months, 12 months, and 24 months)
  We will have patients fill out validated tools for PROs to assess how the patient is doing postoperatively
Oswestry Disability Index (ODI) | 2 years (At baseline, postoperatively at 6 weeks, 3 months, 6 months, 12 months, and 24 months)
  We will have patients fill out validated tools for PROs to assess how the patient is doing postoperatively
Short form survey-12 | 2 years (At baseline, postoperatively at 6 weeks, 3 months, 6 months, 12 months, and 24 months)
  We will have patients fill out validated tools for PROs to assess how the patient is doing postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Agarwal, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No